CLINICAL TRIAL: NCT01985360
Title: International Study of Comparative Health Effectiveness With Medical and Invasive Approaches-Chronic Kidney Disease Trial
Brief Title: ISCHEMIA-Chronic Kidney Disease Trial
Acronym: ISCHEMIA-CKD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: New York University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Duke University (Other); Stanford University (Other); Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-01059; U01HL117905 (NIH)
Record Dates: First submitted 2013-11-04; First posted 2013-11-15 (Estimated); Results first posted 2020-09-10 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-09

CONDITIONS: Cardiovascular Diseases; Coronary Artery Disease; Heart Diseases; Myocardial Ischemia; Kidney Disease; End Stage Renal Failure on Dialysis
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease; Heart Diseases; Myocardial Ischemia; Kidney Diseases | interventions — Cardiac Catheterization; Coronary Artery Bypass; Percutaneous Coronary Intervention; Dosage Forms; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Invasive Strategy (INV) (Active Comparator): Routine invasive strategy with cardiac catheterization followed by revascularization (Percutaneous Coronary Intervention or Coronary Artery Bypass Graft Surgery) plus optimal medical therapy.
  Interventions: Procedure: Cardiac Catheterization; Procedure: Coronary Artery Bypass Graft Surgery; Procedure: Percutaneous Coronary Intervention; Behavioral: Lifestyle; Drug: Medication
- Conservative Strategy (CON) (Active Comparator): Optimal medical therapy with cardiac catheterization and revascularization reserved for patients with OMT failure.
  Interventions: Behavioral: Lifestyle; Drug: Medication

INTERVENTIONS:
Procedure: Cardiac Catheterization — Narrowed blood vessels can be opened without surgery using stents or can be bypassed with surgery. To determine which is the best approach for you the doctor needs to look at your blood vessels to see where the narrowings are and how much narrowing there is. This is done by a procedure known as a cardiac catheterization.
  Other Names: cath
  Arms: Invasive Strategy (INV)
Procedure: Coronary Artery Bypass Graft Surgery — Artery narrowing is bypassed during surgery with a healthy artery or vein from another part of the body. This is known as coronary artery bypass grafting, or CABG (said "cabbage"). The surgery creates new routes around narrowed and blocked heart arteries. This allows more blood flow to the heart.
  Other Names: CABG
  Arms: Invasive Strategy (INV)
Procedure: Percutaneous Coronary Intervention — Percutaneous coronary intervention may be done as part of the cardiac catheterization procedure. With this procedure a small, hollow, mesh tube (stent) is inserted into the narrowed part of the artery. The stent pushes the plaque against the artery wall, and opens the vessel to allow better blood flow.
  Other Names: PCI
  Arms: Invasive Strategy (INV)
Behavioral: Lifestyle — Diet, physical activity, smoking cessation
  Other Names: Behavior change
Drug: Medication — antiplatelet, statin, other lipid lowering, antihypertensive, and anti-ischemic medical therapies
  Other Names: Pharmacologic Therapy

SUMMARY:
The purpose of the ISCHEMIA-CKD trial is to determine the best management strategy for patients with stable ischemic heart disease (SIHD), at least moderate inducible ischemia and advanced chronic kidney disease (CKD; estimated glomerular filtration rate [eGFR] <30 ml/min/1.73 m² or on dialysis). This is a multicenter randomized controlled trial of 777 randomized participants with advanced CKD. Participants were assigned at random to a routine invasive strategy (INV) with cardiac catheterization (cath) followed by revascularization (if suitable) plus optimal medical therapy (OMT) or to a conservative strategy (CON) of OMT, with cath and revascularization reserved for those who fail OMT. The trial is designed to run seamlessly in parallel to the main ISCHEMIA trial as a companion trial.

SPECIFIC AIMS

A. Primary Aim. The primary aim of the ISCHEMIA-CKD trial is to determine whether an invasive strategy of cardiac cath followed by optimal revascularization, in addition to OMT, will reduce the primary composite endpoint of death or nonfatal myocardial infarction in participants with SIHD and advanced CKD over an average follow-up of approximately 2.8 years compared with an initial conservative strategy of OMT alone with catheterization reserved for those who fail OMT. The primary endpoint is time to centrally adjudicated death or nonfatal myocardial infarction (MI).

B. Secondary Aims. Major: To compare the incident of the composite of death, nonfatal MI, resuscitated cardiac arrest, or hospitalization for unstable angina or heart failure, and angina symptoms and quality of life, as assessed by the Seattle Angina Questionnaire, between the INV and CON strategies. Other secondary aims include: comparing the incidence of the composite of death, nonfatal MI, hospitalization for unstable angina, hospitalization for heart failure, resuscitated cardiac arrest, or stroke; composite of death, nonfatal MI, or stroke; composite endpoints incorporating cardiovascular death; composite endpoints incorporating other definitions of MI as defined in the clinical event charter; individual components of the primary and major secondary endpoints; stroke and health resource utilization, costs, and cost effectiveness.

A major secondary aim of ISCHEMIA-CKD trial is to compare the quality of life (QOL) outcomes-patients' symptoms, functioning and well-being-between those assigned to an invasive strategy as compared with a conservative strategy. In the protocol, angina frequency and disease-specific quality of life measured by the Seattle Angina Questionnaire (SAQ) Angina Frequency and Quality of Life scales, respectively, are described as the tools that will be used to make this comparative assessment. Recent work has indicated that it is possible to combine the information from the individual domain scores in the SAQ into a new Summary Score that captures the information from the SAQ Angina Frequency, Physical Limitation and Quality of Life scales into a single overall score. The advantages of using a summary score as the primary measure of QOL effects of a therapy are a single primary endpoint comparison rather than two or three (eliminating concerns some may have about multiple comparisons) and a more intuitive holistic (patient-centric) interpretation of the effectiveness results. With these advantages in mind, the ISCHEMIA leadership has agreed that the SAQ Summary Score will be designated as the primary way this secondary endpoint will be analyzed and interpreted, with the individual SAQ scores being used in a secondary, explanatory and descriptive role. A key subgroup analysis will be to stratify the results among those with daily/weekly angina (baseline SAQ Angina Frequency score ≤60), monthly angina (SAQ Angina Frequency score 61-99) and no angina (SAQ Angina Frequency score = 100).

Condition: Coronary Disease Procedure: Cardiac catheterization Phase: Phase III Condition: Cardiovascular Diseases Procedure: Angioplasty, Transluminal, Percutaneous Coronary, other catheter-based interventions Phase: Phase III Condition: Heart Diseases Procedure: Coronary Artery Bypass Surgery Phase: Phase III

DETAILED DESCRIPTION:
BACKGROUND:

Among patients with advanced CKD, cardiovascular disease is the leading cause of death,15-30 times higher than the age-adjusted cardiovascular mortality rate in the general population. The projected 4-year mortality is >50% in patients with advanced CKD and is worse than that for patients in the general population who have cancers, heart failure, stroke or MI. Participants with advanced CKD are 5-10 times more likely to die than to reach end stage renal disease (ESRD). Despite this, ~80% of contemporary coronary artery disease (CAD) trials exclude participants with advanced CKD. Most of the treatments aimed at reducing cardiovascular events in advanced CKD are therefore extrapolated from cohorts without advanced CKD. Participants with advanced CKD and cardiovascular disease are undertreated with less frequent use of statins and revascularization therapies, and the optimal management approach to these patients is unknown. Participants with advanced CKD are notably underrepresented in contemporary trials comparing revascularization with medical therapy in SIHD patients, such as the Bypass Angioplasty Revascularization Investigation 2 Diabetes (BARI 2D) trial or the Clinical Outcomes Utilizing Revascularization and Aggressive Drug Evaluation (COURAGE) trial,making any assessment about the efficacy of revascularization plus medical therapy vs. initial medical therapy alone in this cohort problematic.

Participants with advanced CKD are at increased risk for complications of the assigned invasive procedure, specifically contrast-induced acute kidney injury (AKI), dialysis, major bleeding and short-term risk of death. However, there is controversy in the medical literature regarding the incidence (<1% to >30%), effective treatment (saline hydration, N-acetyl cysteine, or sodium bicarbonate), and prognosis of contrast induced AKI (<0.5% to >5% requiring dialysis). In addition, although contrast induced AKI have been associated with increase in short-term mortality, residual confounding in these studies makes interpretation difficulty. Moreover, it is unknown if these short-term increased risks are offset by long-term benefits. Limited observational studies in the CKD cohort suggest a long-term survival benefit of revascularization when compared with medical therapy alone, despite an increase in short-term risks. However, the medical therapy in these trials was not optimized, drug eluting stents were rarely used and there is undoubtedly inherent selection and ascertainment bias with observational studies. The above has resulted in clinical equipoise in the management of these patients, with the rates of revascularization only around 10-45%. The results of ISCHEMIA-CKD will have profound implications for guidelines, health policy, and clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* At least moderate ischemia on an exercise or pharmacologic stress test
* End-stage renal disease on dialysis or estimated glomerular filtration rate (eGFR) <30mL/min/1.73m²
* Willingness to comply with all aspects of the protocol, including adherence to the assigned strategy, medical therapy and follow-up visits
* Willingness to give written informed consent
* Age ≥ 21 years

Exclusion Criteria:

* Left Ventricular Ejection Fraction < 35%
* History of unprotected left main stenosis >50% on prior coronary computed tomography angiography (CCTA) or prior cardiac catheterization (if available)
* Finding of "no obstructive coronary artery disease" (<50% stenosis in all major epicardial vessels) on prior CCTA or prior catheterization, performed within 12 months
* Coronary anatomy unsuitable for either percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG)
* Unacceptable level of angina despite maximal medical therapy
* Very dissatisfied with medical management of angina
* History of noncompliance with medical therapy
* Acute coronary syndrome within the previous 2 months
* PCI within the previous 12 months
* Stroke within the previous 6 months or spontaneous intracranial hemorrhage at any time
* History of ventricular tachycardia requiring therapy for termination, or symptomatic sustained ventricular tachycardia not due to a transient reversible cause
* NYHA class III-IV heart failure at entry or hospitalization for exacerbation of chronic heart failure within the previous 6 months
* Non-ischemic dilated or hypertrophic cardiomyopathy
* Severe valvular disease or valvular disease likely to require surgery or percutaneous valve replacement during the trial
* Allergy to radiographic contrast that cannot be adequately pre-medicated, or any prior anaphylaxis to radiographic contrast
* Planned major surgery necessitating interruption of dual antiplatelet therapy (note that patients may be eligible after planned surgery)
* Life expectancy less than the duration of the trial due to non-cardiovascular comorbidity
* Pregnancy
* High likelihood of significant unprotected left main stenosis, in the judgment of the patient's physician
* Enrollment in a competing trial that involves a non-approved cardiac drug or device
* Inability to comply with the protocol
* Body weight or size exceeding the limit for cardiac catheterization at the site
* Canadian Cardiovascular Society Class III angina of recent onset, OR angina of any class with a rapidly progressive or accelerating pattern
* Canadian Cardiovascular Society Class IV angina, including unprovoked rest angina
* High risk of bleeding which would contraindicate the use of dual antiplatelet therapy
* Cardiac transplant recipient
* Prior CABG, unless CABG was performed more than 12 months ago, and coronary anatomy has been demonstrated to be suitable for PCI or repeat CABG to accomplish complete revascularization of ischemic areas

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 777 (Actual)
Dates: Start 2014-01; Primary Completion 2019-06 (Actual); Study Completion 2020-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harmony Reynolds, MD, MHA, Principal Investigator — NYU Langone Health; Judith Hochman, MD, Study Chair — ISCHEMIA trial Chair, New York University School of Medicine; David Maron, MD, Study Chair — ISCHEMIA trial Co-chair, Stanford University
Locations (1):
- NYU Langone Medical Center, New York, New York, United States

REFERENCES:
- [Background] Bangalore S, Maron DJ, Fleg JL, O'Brien SM, Herzog CA, Stone GW, Mark DB, Spertus JA, Alexander KP, Sidhu MS, Chertow GM, Boden WE, Hochman JS; ISCHEMIA-CKD Research Group. International Study of Comparative Health Effectiveness with Medical and Invasive Approaches-Chronic Kidney Disease (ISCHEMIA-CKD): Rationale and design. Am Heart J. 2018 Nov;205:42-52. doi: 10.1016/j.ahj.2018.07.023. Epub 2018 Aug 1. PMID 30172098
- [Background] Bangalore S, Fayyad R, Hovingh GK, Laskey R, Vogt L, DeMicco DA, Waters DD; Treating to New Targets Steering Committee and Investigators. Statin and the risk of renal-related serious adverse events: Analysis from the IDEAL, TNT, CARDS, ASPEN, SPARCL, and other placebo-controlled trials. Am J Cardiol. 2014 Jun 15;113(12):2018-20. doi: 10.1016/j.amjcard.2014.03.046. Epub 2014 Apr 3. PMID 24793673
- [Background] Bangalore S, Maron DJ, Hochman JS. Evidence-Based Management of Stable Ischemic Heart Disease: Challenges and Confusion. JAMA. 2015 Nov 10;314(18):1917-8. doi: 10.1001/jama.2015.11219. No abstract available. PMID 26547460
- [Background] Stone GW, Hochman JS, Williams DO, Boden WE, Ferguson TB Jr, Harrington RA, Maron DJ. Medical Therapy With Versus Without Revascularization in Stable Patients With Moderate and Severe Ischemia: The Case for Community Equipoise. J Am Coll Cardiol. 2016 Jan 5;67(1):81-99. doi: 10.1016/j.jacc.2015.09.056. Epub 2015 Nov 23. PMID 26616030
- [Background] Bangalore S. Diagnostic, Therapeutic, and Clinical Trial Conundrum of Patients With Chronic Kidney Disease. JACC Cardiovasc Interv. 2016 Oct 24;9(20):2110-2112. doi: 10.1016/j.jcin.2016.08.031. Epub 2016 Sep 28. No abstract available. PMID 27692819
- [Background] Shroff GR, Herzog CA. Coronary Revascularization in Patients with CKD Stage 5D: Pragmatic Considerations. J Am Soc Nephrol. 2016 Dec;27(12):3521-3529. doi: 10.1681/ASN.2016030345. Epub 2016 Aug 4. PMID 27493258
- [Background] Mathew RO, Bangalore S, Lavelle MP, Pellikka PA, Sidhu MS, Boden WE, Asif A. Diagnosis and management of atherosclerotic cardiovascular disease in chronic kidney disease: a review. Kidney Int. 2017 Apr;91(4):797-807. doi: 10.1016/j.kint.2016.09.049. Epub 2016 Dec 28. PMID 28040264
- [Background] Pandya B, Chalhoub JM, Parikh V, Gaddam S, Spagnola J, El-Sayegh S, Bogin M, Kandov R, Lafferty J, Bangalore S. Contrast media use in patients with chronic kidney disease undergoing coronary angiography: A systematic review and meta-analysis of randomized trials. Int J Cardiol. 2017 Feb 1;228:137-144. doi: 10.1016/j.ijcard.2016.11.170. Epub 2016 Nov 9. PMID 27863354
- [Background] Patel AV, Bangalore S. Challenges with Evidence-Based Management of Stable Ischemic Heart Disease. Curr Cardiol Rep. 2017 Feb;19(2):11. doi: 10.1007/s11886-017-0820-7. PMID 28185167
- [Background] Bangalore S, Briguori C. Preventive Strategies for Contrast-Induced Acute Kidney Injury: And the Winner Is.... Circ Cardiovasc Interv. 2017 May;10(5):e005262. doi: 10.1161/CIRCINTERVENTIONS.117.005262. No abstract available. PMID 28487357
- [Background] Mathew RO, Bangalore S, Sidhu MS, Fleg JL, Maddux FW. Increasing inclusion of patients with advanced chronic kidney disease in cardiovascular clinical trials. Kidney Int. 2018 Apr;93(4):787-788. doi: 10.1016/j.kint.2017.11.028. No abstract available. PMID 29571453
- [Background] Chaudhry RI, Mathew RO, Sidhu MS, Sidhu-Adler P, Lyubarova R, Rangaswami J, Salman L, Asif A, Fleg JL, McCullough PA, Maddux F, Bangalore S. Detection of Atherosclerotic Cardiovascular Disease in Patients with Advanced Chronic Kidney Disease in the Cardiology and Nephrology Communities. Cardiorenal Med. 2018;8(4):285-295. doi: 10.1159/000490768. Epub 2018 Aug 3. PMID 30078001
- [Background] Bangalore S, Guo Y, Samadashvili Z, Blecker S, Xu J, Hannan EL. Revascularization in Patients With Multivessel Coronary Artery Disease and Chronic Kidney Disease: Everolimus-Eluting Stents Versus Coronary Artery Bypass Graft Surgery. J Am Coll Cardiol. 2015 Sep 15;66(11):1209-1220. doi: 10.1016/j.jacc.2015.06.1334. PMID 26361150
- [Background] Bangalore S. Stress testing in patients with chronic kidney disease: The need for ancillary markers for effective risk stratification and prognosis. J Nucl Cardiol. 2016 Jun;23(3):570-4. doi: 10.1007/s12350-015-0264-7. Epub 2015 Aug 22. No abstract available. PMID 26297196
- [Background] Patel A, Bangalore S. Revascularization Strategies in Chronic Kidney Disease: Percutaneous Coronary Intervention vs. Coronary Artery Bypass Graft Surgery. Janani Rangaswami, Dr. Edgar V. Lerman, and Dr. Claudio Ronco (Eds), Cardio-nephrology: Confluence of the Heart and Kidney in Clinical Practice. London: Springer-Verlag
- [Derived] Sidhu MS, Alexander KP, Huang Z, Mathew RO, Newman JD, O'Brien SM, Pellikka PA, Lyubarova R, Bockeria O, Briguori C, Kretov EL, Mazurek T, Orso F, Roik MF, Sajeev C, Shutov EV, Rockhold FW, Borrego D, Balter S, Stone GW, Chaitman BR, Goodman SG, Fleg JL, Reynolds HR, Maron DJ, Hochman JS, Bangalore S; ISCHEMIA-CKD Research Group. Cause-Specific Mortality in Patients With Advanced Chronic Kidney Disease in the ISCHEMIA-CKD Trial. JACC Cardiovasc Interv. 2023 Jan 23;16(2):209-218. doi: 10.1016/j.jcin.2022.10.062. PMID 36697158
- [Derived] Mathew RO, Maron DJ, Anthopolos R, Fleg JL, O'Brien SM, Rockhold FW, Briguori C, Roik MF, Mazurek T, Demkow M, Malecki R, Ye Z, Kaul U, Miglinas M, Stone GW, Wald R, Charytan DM, Sidhu MS, Hochman JS, Bangalore S. Guideline-Directed Medical Therapy Attainment and Outcomes in Dialysis-Requiring Versus Nondialysis Chronic Kidney Disease in the ISCHEMIA-CKD Trial. Circ Cardiovasc Qual Outcomes. 2022 Oct;15(10):e008995. doi: 10.1161/CIRCOUTCOMES.122.008995. Epub 2022 Oct 4. PMID 36193750
- [Derived] Chaitman BR, Cyr DD, Alexander KP, Pracon R, Bainey KR, Mathew A, Acharya A, Kunichoff DF, Fleg JL, Lopes RD, Sidhu MS, Anthopolos R, Rockhold FW, Stone GW, Maron DJ, Hochman JS, Bangalore S. Cardiovascular and Renal Implications of Myocardial Infarction in the ISCHEMIA-CKD Trial. Circ Cardiovasc Interv. 2022 Aug;15(8):e012103. doi: 10.1161/CIRCINTERVENTIONS.122.012103. Epub 2022 Aug 16. PMID 35973009
- [Derived] Briguori C, Mathew RO, Huang Z, Mavromatis K, Hickson LJ, Lau WL, Mathew A, Mahajan S, Wheeler DC, Claes KJ, Chen G, Nolasco FEB, Stone GW, Fleg JL, Sidhu MS, Rockhold FW, Chertow GM, Hochman JS, Maron DJ, Bangalore S. Dialysis Initiation in Patients With Chronic Coronary Disease and Advanced Chronic Kidney Disease in ISCHEMIA-CKD. J Am Heart Assoc. 2022 Mar 15;11(6):e022003. doi: 10.1161/JAHA.121.022003. Epub 2022 Mar 9. PMID 35261290
- [Derived] Herzog CA, Simegn MA, Xu Y, Costa SP, Mathew RO, El-Hajjar MC, Gulati S, Maldonado RA, Daugas E, Madero M, Fleg JL, Anthopolos R, Stone GW, Sidhu MS, Maron DJ, Hochman JS, Bangalore S. Kidney Transplant List Status and Outcomes in the ISCHEMIA-CKD Trial. J Am Coll Cardiol. 2021 Jul 27;78(4):348-361. doi: 10.1016/j.jacc.2021.05.001. Epub 2021 May 11. PMID 33989711
- [Derived] Bangalore S, Maron DJ, O'Brien SM, Fleg JL, Kretov EI, Briguori C, Kaul U, Reynolds HR, Mazurek T, Sidhu MS, Berger JS, Mathew RO, Bockeria O, Broderick S, Pracon R, Herzog CA, Huang Z, Stone GW, Boden WE, Newman JD, Ali ZA, Mark DB, Spertus JA, Alexander KP, Chaitman BR, Chertow GM, Hochman JS; ISCHEMIA-CKD Research Group. Management of Coronary Disease in Patients with Advanced Kidney Disease. N Engl J Med. 2020 Apr 23;382(17):1608-1618. doi: 10.1056/NEJMoa1915925. Epub 2020 Mar 30. PMID 32227756
- [Derived] Spertus JA, Jones PG, Maron DJ, Mark DB, O'Brien SM, Fleg JL, Reynolds HR, Stone GW, Sidhu MS, Chaitman BR, Chertow GM, Hochman JS, Bangalore S; ISCHEMIA-CKD Research Group. Health Status after Invasive or Conservative Care in Coronary and Advanced Kidney Disease. N Engl J Med. 2020 Apr 23;382(17):1619-1628. doi: 10.1056/NEJMoa1916374. Epub 2020 Mar 30. PMID 32227754
- See also: Official website of the ISCHEMIA Trial — http://www.ischemiatrial.org
- See also: Official website of the ISCHEMIA-CKD Trial — http://ischemiackd.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Invasive Strategy (INV): Routine invasive strategy with cardiac catheterization followed by revascularization + optimal medical therapy.
  * Cardiac Catheterization: Narrowed blood vessels can be opened without surgery using stents or bypassed with surgery. The doctor will examine blood vessels to determine the location and extent of narrowings.
  * Coronary Artery Bypass Graft Surgery (CABG): Artery narrowing is bypassed during surgery with a healthy artery or vein from another part of the body. This creates new routes around narrowed/blocked heart arteries.
  * Percutaneous Coronary Intervention: A small, hollow, mesh tube (stent) is inserted into the narrowed part of the artery. The stent pushes the plaque against the artery wall, and opens the vessel to allow better blood flow.
  Lifestyle: Diet, physical activity, smoking cessation Medication: antiplatelet, statin, other lipid lowering, antihypertensive, and anti-ischemic medical therapies
Period: Overall Study
Arm/Group | Invasive Strategy (INV) | Conservative Strategy (CON)
Started | 388 | 389
Completed | 379 | 386
Not Completed | 9 | 3
Not completed — Withdrawal by Subject | 4 | 0
Not completed — Lost to Follow-up | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Invasive Strategy (INV) | Conservative Strategy (CON) | Total
Number analyzed (Participants) | 388 | 389 | 777
Age, Continuous [Mean (Full Range); unit: years] | 62 [55 to 69] | 64 [56 to 70] | 63 [55 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 122 | 242
  Male | 268 | 267 | 535
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 54 | 44 | 98
  Not Hispanic or Latino | 318 | 319 | 637
  Unknown or Not Reported | 16 | 26 | 42
Region of Enrollment [Number; unit: participants]
  North America | 95 | 88 | 183
  Europe | 120 | 119 | 239
  Africa | 1 | 2 | 3
  Pacifica | 3 | 7 | 10
  Middle East | 3 | 3 | 6
  South America | 27 | 22 | 49

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Death From Any Cause or Myocardial Infarction
Time Frame: 2.2 years
Measure: Count of Participants; unit: Participants
Groups:
- Invasive Strategy: Invasive Strategy
- Conservative Strategy: Conservative Strategy
Arm/Group | Invasive Strategy | Conservative Strategy
Number analyzed (Participants) | 388 | 389
Participants | 123 | 129

2. Primary Outcome: Cumulative Event Rate of Death From Any Cause or Myocardial Infarction
Description: This measure represents the estimated cumulative probability of experiencing Death from any cause or Myocardial Infarction within the indicated timeframe in each treatment group. The interpretation of the measure is similar to Kaplan-Meier event rates. Estimates are expressed as percentages ranging from 0% (endpoint is certain not to occur) to 100% (endpoint is certain to occur).
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: cumulative event rate - %
Arm/Group | Invasive Strategy | Conservative Strategy
Number analyzed (Participants) | 388 | 389
cumulative event rate - % | 36.4 [30.5 to 42.2] | 36.7 [31.1 to 42.4]
Statistical Analysis 1: Comparison: Invasive Strategy vs Conservative Strategy; Test type: Other; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.79 to 1.29]

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Invasive Strategy | Conservative Strategy
All-Cause Mortality (participants affected / at risk) | 94/388 | 98/389
Serious Adverse Events (participants affected / at risk) | 75/388 | 61/389
Other Adverse Events (participants affected / at risk) | 0/388 | 0/389
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Invasive Strategy (N=388) | Conservative Strategy (N=389)
Death from any cause or Initiation of dialysis (Renal and urinary disorders) | 75 (75) | 61 (61) — This category consists of patients who were not receiving dialysis at baseline

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-18): https://cdn.clinicaltrials.gov/large-docs/60/NCT01985360/Prot_SAP_000.pdf